CLINICAL TRIAL: NCT02769715
Title: Laser-sintered Removable Partial Dentures: a Crossover Pilot Clinical Trial
Brief Title: A Study About Patient Satisfaction With Laser-sintered Removable Partial Dentures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faleh Tamimi (Other)
Collaborators: 3DRPD Inc. (Industry)
Responsible Party: Sponsor-Investigator, Faleh Tamimi, Assistant Professor and Canada Research Chair in Translational Craniofacial Research, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 12-452 BMD
Record Dates: First submitted 2016-04-22; First posted 2016-05-12 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Partially Edentulous Jaws
Keywords: Removable partial dentures; partial edentulism

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cast removable partial denture (Active Comparator): patients received cast removable partial dentures fabricated using traditional lost-wax casting technique.
  Interventions: Other: cast removable partial dentures
- laser-sintered removable partial denture (Experimental): patients received removable partial dentures fabricated using laser-sintering.
  Interventions: Device: Laser-sintered removable partial denture

INTERVENTIONS:
Device: Laser-sintered removable partial denture — The master cast was scanned using 3D scanner. In the digital file, the path of insertion was determined using a special software. The survey line was drawn and all undesirable undercuts were eliminated. After that, the entire framework design was built virtually 3 dimensionally using a special software (3Shape Software) according to the specified design in three steps: deciding the contour of the component, building the tissue surface then creating the polished surface. The file was saved in STL file and was transferred to rapid prototyping machine. Framework was produced by selective laser sintering technique using the alloy powder (Sintech Metal).
  Arms: laser-sintered removable partial denture
Other: cast removable partial dentures — The denture was fabricated traditionally using lost-wax casting technique.
  Arms: cast removable partial denture

SUMMARY:
Removable partial dentures (RPDs) are traditionally fabricated by lost-wax casting technique, a time-consuming and very laborious manual technique. Recently, fabricating removable partial dentures using computer designing and laser sintering techniques have been introduced. The purpose of this study was to evaluate the patient satisfaction with new computer-generated removable partial dentures and compare it to the traditional removable partial dentures.

DETAILED DESCRIPTION:
Patients seeking Removable partial dentures in the undergraduate clinic at McGill University were asked to participate in the study. Patients were treated by undergraduate students under the supervision of expert prosthodontists. Both the dentists treating the case and the patients were blinded to the type of RPD used. The Principal investigator was responsible for preparing the laboratory prescriptions and sending the final impressions to the dental lab in order to assure blinding of the patient and the treating dentists.

Patients were treated according to standardized clinical procedures. Both dentures were fabricated from one master cast to ensure standardization. The cast was scanned digitally to fabricate the laser-sintered dentures, and then was used to fabricate the cast dentures traditionally using lost-wax casting technique. For each patient, two dentures were fabricated from one final impression; one by casting technique and the other by laser-sintering. Patients were given randomly one denture first and followed-up for 1, 2 and 4 weeks. Then, they were given the second denture and followed-up again. At each follow-up visit, patients filled McGill Denture Satisfaction Instrument. At the end of the study patients were asked which denture they prefer to keep.

ELIGIBILITY:
Inclusion Criteria:

* partially edentulous
* have adequate space for regularly sized prosthetic teeth and metal frame(s)
* be able to maintain adequate oral hygiene and clean their dentures; do not have major systemic health problems that could interfere with general oral health
* have an adequate understanding of written and spoken English or French
* be capable of giving written informed consent and fill out questionnaires

Exclusion Criteria:

* there is a lack of minimum interocclusal space to accommodate a metal frame and acrylic material
* they have acute or chronic symptoms of parafunctional disorders
* they have inflammatory mucosal conditions such as lichen planus, progressive periodontitis or others
* they have a history of radiation therapy to the orofacial region
* there are health conditions that may jeopardize the treatment, such as alcoholism,
* they are taking any phenytoin (Dilantin), cortisone or insulin
* they have a severe/serious illness that requires frequent hospitalization
* they have impaired cognitive or motor function
* they are unable to return for evaluations/study recalls

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-01; Primary Completion 2015-06 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Mean of patient satisfaction measured by McGill Denture Satisfaction Survey using visual analog scale from 0-100 | after 4 weeks
  Mean patient satisfaction in McGill Denture Satisfaction Survey was assessed in regard to 9 aspects of the dentures; general satisfaction, chewing efficiency, chewing ability, easiness to clean, stability, comfort and oral condition. Mean of patient satisfaction in each of these 9 aspects will be presented for both cast and laser-sintered dentures.

SECONDARY OUTCOMES:
Number of participants who choose to keep the laser-sintered removable partial dentures | after 2 months
  Patients will be asked which denture did they prefer to keep after trying both cast and laser-sintered removable partial dentures. The number of patients who preferred each denture will be presented as well as the number of patients who have no preference.

CONTACTS AND LOCATIONS:
Overall Officials: Faleh Tamimi, Principal Investigator — McGill University Faculty of Dentistry; Rubens Albuquerque, Principal Investigator — McGill University Faculty of Dentistry
Locations (1):
- McGill University Faculty of Dentistry, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
The patients' demographic data including (age, sex, the number of missing anterior and posterior teeth, previous denture experience, denture arch, opposing arch and Kennedy classification of the denture, first denture received and preferred denture) will be published in a scientific journal without any indication of personal identity of the patients.

REFERENCES:
- [Background] Koutsoukis T, Zinelis S, Eliades G, Al-Wazzan K, Rifaiy MA, Al Jabbari YS. Selective Laser Melting Technique of Co-Cr Dental Alloys: A Review of Structure and Properties and Comparative Analysis with Other Available Techniques. J Prosthodont. 2015 Jun;24(4):303-12. doi: 10.1111/jopr.12268. PMID 26129918
- [Background] Lima JM, Anami LC, Araujo RM, Pavanelli CA. Removable partial dentures: use of rapid prototyping. J Prosthodont. 2014 Oct;23(7):588-91. doi: 10.1111/jopr.12154. Epub 2014 Apr 18. PMID 24750472
- [Background] Williams RJ, Bibb R, Eggbeer D, Collis J. Use of CAD/CAM technology to fabricate a removable partial denture framework. J Prosthet Dent. 2006 Aug;96(2):96-9. doi: 10.1016/j.prosdent.2006.05.029. PMID 16911885
- [Derived] Almufleh B, Emami E, Alageel O, de Melo F, Seng F, Caron E, Nader SA, Al-Hashedi A, Albuquerque R, Feine J, Tamimi F. Patient satisfaction with laser-sintered removable partial dentures: A crossover pilot clinical trial. J Prosthet Dent. 2018 Apr;119(4):560-567.e1. doi: 10.1016/j.prosdent.2017.04.021. Epub 2017 Jul 11. PMID 28709680